CLINICAL TRIAL: NCT00771485
Title: Study of Efficacy of Bowel Preparation Before Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C.B. Fleet Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PL08.01
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Bowel Cleansing Prior to Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: FM-602
- 2 (Other)
  Interventions: Drug: Marketed Bowel Cleanser

INTERVENTIONS:
Drug: FM-602 — Study of Efficacy of Bowel Preparation Before Colonoscopy
  Arms: 1
Drug: Marketed Bowel Cleanser — Marketed bowel cleanser
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of FM-602 as a bowel preparation before colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Are men or nonpregnant women who are scheduled for an elective colonoscopy and who are at least 18 years of age,
* Are, in the opinion of the Investigator, able to communicate with study personnel and comply with the requirements of the study,
* Are able and willing to follow the study-specified testing including the diet and hydration regimen, and
* Have been informed of the nature and risks of the study and have given written informed consent at Screening and before any study-related tests are done.

Exclusion Criteria:

* Have any known contraindications to the study procedures or treatment,
* Have clinically significant active cardiovascular disease, including a history of myocardial infarction, within the past 6 months and/or heart failure
* Have known or suspected electrolyte abnormalities, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon, or ileus,
* Have any history of prior colon surgery,
* History of active inflammatory bowel disease,
* Have clinical evidence of dehydration,
* Are pregnant or breast-feeding,
* Are unwilling to abstain from alcohol consumption from the day before colonoscopy until discharged from the study,
* Are unwilling to use any prohibited medications, including laxatives, 4 days before receiving the first study dose,
* Have received any investigational agent within 30 days before dosing,
* Have any known or suspected allergies, sensitivity or an unwillingness to consume components of the study medication,
* Known or suspected phenylketonuria (PKU) or sensitivity to products containing phenylalanine, or is on a phenylalanine-reduced diet,
* A history of hemolysis or taking concomitant medications known to precipitate hemolytic reactions,
* Have any other condition which in the Investigator's opinion would make the subject unsuitable for inclusion into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of bowel cleansing assessed by the examining physician | During colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sherrie McNamara, RN, MSN, MBA, Study Director — C.B. Fleet Company, Inc.
Locations (3):
- United States (3):
  - Advanced Clinical Research Institute, Anaheim, California
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia